CLINICAL TRIAL: NCT01310062
Title: Strategic Alliance for The Development of Diagnostic Biomarker Panels for Hepatitis and Liver Cancer
Brief Title: The Development of Diagnostic Biomarker Panels for Hepatitis and Liver Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ministry of Health, Malaysia (Other Government)
Collaborators: GeneNews Sdn Bhd (Unknown)
Responsible Party: Professor Dato' Dr. Liew Choong Chin, GeneNews Sdn Bhd
Other Study IDs: 09-317-3991
Record Dates: First submitted 2011-03-04; First posted 2011-03-07 (Estimated); Last update posted 2011-03-07 (Estimated); Status verified 2011-03

CONDITIONS: Hepatitis B,Chronic; Carcinoma,Hepatocellular
Keywords: hepatocellular carcinoma; microarray; gene expression profiling; biomarkers
MeSH Terms: conditions — Hepatitis B, Chronic; Carcinoma, Hepatocellular

STUDY DESIGN:
Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Red blood cell and white blood cell
Oversight: Data Monitoring Committee: No

SUMMARY:
More recent studies have shown that the HBV-infected population has a greater risk of development of hepatocellular carcinoma. Nevertheless, there are still a significant number of people chronically infected by HBV who do not develop the complication. Hence, there exist biological markers that could be indicator for the disease-inducing and carcinogenic potential of the virus.

ELIGIBILITY:
Inclusion Criteria:

* Patients of at least 21 years old on day of giving consent for study
* Patients must be able and wiling to give an informed consent
* Patient with chronic HBV infection
* Patient with active hepatocellular carcinoma and chronic hepatitis B
* Healthy subjects

Exclusion Criteria:

* Patients who have co-infection with HIV or chronic hepatitis C
* Subjects with other types of cancer

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Selected hospitals for study
Sampling Method: Non-Probability Sample
Enrollment: 1600 (Estimated)
Dates: Start 2010-08; Study Completion 2012-08 (Estimated)

CONTACTS AND LOCATIONS:
Locations (8):
- Malaysia (8):
  - Sultanah Bahiyah Hospital, Alor Star, Kedah
  - Kuala Lumpur Hospital, Kuala Lumpur, Kuala Lumpur
  - Island Hospital, Pulau Pinang, Pulau Pinang
  - Lam Wah Ee Hospital, Pulau Pinang, Pulau Pinang
  - Penang Hospital, Pulau Pinang, Pulau Pinang
  - Queen Elizabeth Hospital, Kota Kinabalu, Sabah
  - Hospital Umum Kuching Sarawak, Kuching, Sarawak
  - Selayang Hospital, Selayang Baru Utara, Selangor